CLINICAL TRIAL: NCT00082537
Title: A Multicenter, Double-Blind, Randomized, Comparative Study to Evaluate the Safety, Tolerability, and Efficacy of Caspofungin Versus (Amphotericin B) Liposome for Injection as Empirical Therapy in Pediatric Patients With Persistent Fever and Neutropenia
Brief Title: MK0991 Versus Amphotericin B for Empirical Therapy in Febrile, Neutropenic Pediatric Patients (0991-044)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0991-044; Formerly-0404ETPP; MK0991-044; 2004_101
Record Dates: First submitted 2004-05-11; First posted 2004-05-13 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Neutropenia; Fever
MeSH Terms: conditions — Neutropenia; Fever | interventions — Caspofungin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: caspofungin acetate — Duration of Treatment: 28-90 days
  Other Names: MK0991
Drug: Comparator: AmBisome — Duration of Treatment: 28-90 days

SUMMARY:
This study is a double-blind, randomized study of MK0991 versus liposomal amphotericin B in the empirical treatment of pediatric patients (ages 2 through 17 years) who have an absolute neutrophil count (ANC) below 500/microliter and who have fever despite broad antibiotic coverage. Such patients would be candidates for empirical therapy with an intravenous anti-fungal agent.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 2 through 17 years of age
* Absolute Neutrophil Count (ANC) is below 500/microliter
* Have persistent fever (at least 4 days) despite antibiotic therapy

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2004-04; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To estimate the proportion of patients treated with caspofungin reporting one or more clinical and/or laboratory drug-related adverse experience(s) during the study drug therapy period plus 14 days posttherapy

SECONDARY OUTCOMES:
Proportion of patients with a favorable overall response

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Maertens JA, Madero L, Reilly AF, Lehrnbecher T, Groll AH, Jafri HS, Green M, Nania JJ, Bourque MR, Wise BA, Strohmaier KM, Taylor AF, Kartsonis NA, Chow JW, Arndt CA, DePauw BE, Walsh TJ; Caspofungin Pediatric Study Group. A randomized, double-blind, multicenter study of caspofungin versus liposomal amphotericin B for empiric antifungal therapy in pediatric patients with persistent fever and neutropenia. Pediatr Infect Dis J. 2010 May;29(5):415-20. doi: 10.1097/INF.0b013e3181da2171. PMID 20431381
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html